CLINICAL TRIAL: NCT02753400
Title: A Multicenter, Randomized, Double-Masked, Placebo-Controlled, Pilot Study to Evaluate Effects of Emixustat Hydrochloride on Aqueous Humor Biomarkers Associated With Proliferative Diabetic Retinopathy
Brief Title: Study to Evaluate Effects of Emixustat Hydrochloride in Subjects With Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4429-203
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — emixustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emixustat hydrochloride (Experimental): Week 1- Four tablets (2 placebo, 2 emixustat HCl Strength A)
  Week 2- Four tablets (2 placebo, 2 emixustat HCl Strength B)
  Week 3- Four tablets (2 placebo, 2 emixustat HCl Strength C)
  Week 4- Four emixustat HCl tablets (Strength C)
  All tablets are administered orally once daily. After week 4, all subjects will be held at a stable dose for the remainder of the 12-week dosing regimen.
  Interventions: Drug: emixustat hydrochloride; Other: Placebo
- Placebo (Placebo Comparator): Four placebo tablets are administered orally once daily for 12 weeks; Subjects in the placebo group will be mock-titrated on the same schedule as those in the active arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: emixustat hydrochloride — Tablet for oral administration
  Other Names: ACU-4429, Emixustat HCl
  Arms: Emixustat hydrochloride
Other: Placebo — Placebo tablets for oral administration contain only inactive ingredients

SUMMARY:
To evaluate the effects of oral emixustat hydrochloride (emixustat) on aqueous humor biomarkers associated with proliferative diabetic retinopathy (PDR) from baseline to week 12.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-masked, placebo-controlled study to evaluate the effects of emixustat in subjects with PDR. Subjects will be randomly assigned to either emixustat or placebo arms and treated once daily (QD) for 12 weeks. Doses of emixustat will be doubled on a weekly basis until week 4 after which all subjects will be held at a stable dose for the remainder of the 12-week dosing regimen. Subjects in the placebo group will be mock-titrated on the same schedule as those in the emixustat arm.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Documented diagnosis of type 1 or type 2 diabetes mellitus
* Meets specific ocular criteria for the study eye including but not limited to, the presence of PDR with or without diabetic macular edema in study eye for which treatment can be deferred for at least 4 weeks after Day 1 visit
* Media clarity, pupillary dilation, and subject cooperation sufficient to obtain adequate assessments

Exclusion Criteria:

* Any condition that would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease or glycemic control)
* History of myocardial infarction or other acute cardiac event
* History of chronic renal failure requiring dialysis or kidney transplant
* Prior participation in any clinical study of emixustat
* Treatment with any investigational study drug within 30 days of screening
* Known allergy to fluorescein sodium for injection in angiography
* Treatment with specific prohibited medications or therapy beginning 4 weeks prior to screening and throughout the duration of the study
* History of systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization
* Pre-specified laboratory abnormalities at screening
* Specific ocular characteristics in the study eye
* Male subjects who are not surgically sterile and are not willing to practice a medically accepted method of birth control with their female partner of childbearing potential from screening through 30 days following completion of the study
* Female subjects of childbearing potential who are not willing to practice a medically accepted method of birth control with their non-surgically sterile male sexual partner from screening through 30 days following completion of the study
* Female subjects who are pregnant or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Responsible Medical Officer, Study Director — Kubota Vision Inc.
Locations (1):
- Retina Institute of California, Arcadia, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kubota R, Jhaveri C, Koester JM, Gregory JK. Effects of emixustat hydrochloride in patients with proliferative diabetic retinopathy: a randomized, placebo-controlled phase 2 study. Graefes Arch Clin Exp Ophthalmol. 2021 Feb;259(2):369-378. doi: 10.1007/s00417-020-04899-y. Epub 2020 Aug 27. PMID 32852613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from May 2016 through July 2017 at 8 sites in the United States
Groups:
- Emixustat Hydrochloride: Week 1- Four tablets (2 placebo, 2 emixustat HCl Strength A)
  Week 2- Four tablets (2 placebo, 2 emixustat HCl Strength B)
  Week 3- Four tablets (2 placebo, 2 emixustat HCl Strength C)
  Week 4- Four emixustat HCl tablets (Strength C)
  All tablets are administered orally once daily. After week 4, all subjects will be held at a stable dose for the remainder of the 12-week dosing regimen.
  emixustat hydrochloride: Tablet for oral administration
  Placebo: Placebo tablets for oral administration contain only inactive ingredients
Period: Overall Study
Arm/Group | Emixustat Hydrochloride | Placebo
Started | 12 | 12
Completed | 7 | 11
Not Completed | 5 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emixustat Hydrochloride | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (7.06) | 47.4 (11.29) | 49.8 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Aqueous Humor Concentration of the Following Biomarkers:IL-6, IL-8, IP-10, PDGF-AA, TGFβ-1, MCP-1, IL-1β, and VEGF, to be Reported in pg/mL Values
Description: All values for IL-1β were below the lower limit of detection and were recorded as zero. Tests for IP-10 and MCP-1 failed accuracy and stability testing during assay development and were dropped from the study. The assay for PDGF-AA could not be developed.and results were not reported.
Time Frame: Baseline and 12 weeks
Population: Not all subjects had primary endpoint end-of-treatment data.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Emixustat Hydrochloride | Placebo
Number analyzed (Participants) | 12 | 11
pg/ml
  IL-6, change from baseline: number analyzed (Participants) | 9 | 11
  IL-6, change from baseline | 45.6 (137.1) | 4.9 (12.6)
  IL-8, change from baseline: number analyzed (Participants) | 9 | 11
  IL-8, change from baseline | 4.2 (5.1) | 2.6 (4.6)
  TGFβ-1, change from baseline: number analyzed (Participants) | 9 | 11
  TGFβ-1, change from baseline | -19.9 (32.4) | -17.5 (43.7)
  VEGF, change from baseline: number analyzed (Participants) | 9 | 11
  VEGF, change from baseline | -38.0 (115.1) | -24.8 (277.2)

ADVERSE EVENTS:
Time Frame: Day 115
Arm/Group | Emixustat Hydrochloride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/11
Other Adverse Events (participants affected / at risk) | 12/12 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emixustat Hydrochloride (N=12) | Placebo (N=11)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Emixustat Hydrochloride (N=12) | Placebo (N=11)
DELAYED DARK ADAPTATION (Eye disorders) | 9 | 1
BLINDNESS DAY (Eye disorders) | 4 | 3
VISION BLURRED (Eye disorders) | 1 | 6
VISUAL IMPAIRMENT (Eye disorders) | 6 | 1
VITREOUS FLOATERS (Eye disorders) | 4 | 2
VISUAL ACUITY REDUCED (Eye disorders) | 4 | 1
CHROMATOPSIA (Eye disorders) | 4 | 0
VISUAL ACUITY TESTS ABNORMAL (Investigations) | 2 | 2
VITREOUS HAEMORRHAGE (Eye disorders) | 3 | 1
DIABETIC RETINAL OEDEMA (Eye disorders) | 1 | 2
ERYTHROPSIA (Eye disorders) | 3 | 0
HEADACHE (Nervous system disorders) | 2 | 1
PHOTOPHOBIA (Eye disorders) | 1 | 2
RETINAL NEOVASCULARISATION (Eye disorders) | 1 | 2
RETINAL ANEURYSM (Eye disorders) | 2 | 0
RETINAL DETACHMENT (Eye disorders) | 2 | 0
RETINAL EXUDATES (Eye disorders) | 0 | 2
RETINAL HAEMORRHAGE (Eye disorders) | 1 | 1
VITREOUS DETACHMENT (Eye disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 1 | 0
BRONCHITIS VIRAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CATARACT (Eye disorders) | 0 | 1
CATARACT CORTICAL (Eye disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
DIABETIC RETINOPATHY (Eye disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1
EYE IRRITATION (Eye disorders) | 0 | 1
EYE PAIN (Eye disorders) | 0 | 1
EYE PRURITUS (Eye disorders) | 0 | 1
FATIGUE (General disorders) | 0 | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 0
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 0 | 1
HAEMATOCRIT DECREASED (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
HOT FLUSH (Vascular disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
HYPOTHYROIDISM (Metabolism and nutrition disorders) | 1 | 0
LIGAMENT SPRAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
MACULAR FIBROSIS (Eye disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
NIGHT BLINDNESS (Eye disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1
PUNCTATE KERATITIS (Eye disorders) | 0 | 1
RETINAL CYST (Eye disorders) | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 1
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
VISUAL BRIGHTNESS (Eye disorders) | 0 | 1
VITREOUS ADHESIONS (Eye disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
WEIGHT INCREASED (Investigations) | 1 | 0
XANTHOPSIA (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT02753400/Prot_SAP_000.pdf